CLINICAL TRIAL: NCT02997761
Title: A Phase 2 Study of Ibrutinib and Blinatumomab in Relapsed and Refractory B-Cell Acute Lymphoblastic Leukemia
Brief Title: Ibrutinib and Blinatumomab in Treating Patients With Relapsed or Refractory B Acute Lymphoblastic Leukemia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Brian Jonas (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Pharmacyclics LLC. (Industry)
Responsible Party: Sponsor-Investigator, Brian Jonas, Principal Investigator, University of California, Davis
Organization: University of California, Davis (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 945122; UCDCC#266 (Other: UC Davis IRB); UCDCC#266 (Other: University of California Davis Comprehensive Cancer Center); P30CA093373 (NIH); NCI-2016-01882 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2016-12-12; First posted 2016-12-20 (Estimated); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Adult B Acute Lymphoblastic Leukemia; Philadelphia Chromosome Positive
MeSH Terms: conditions — Burkitt Lymphoma | interventions — blinatumomab; N,N-dicyclohexyl-isoborneol-10-sulfonamide; ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (ibrutinib, blinatumomab) (Experimental): INDUCTION THERAPY: Patients receive ibrutinib PO QD on days 1-49 of course 1 and days 1-42 of course 2, and blinatumomab IV on days 8-35 of course 1 and days 1-28 of course 2 in the absence of disease progression or unacceptable toxicity.
  CONSOLIDATION THERAPY: Patients with CR/CRi after Induction Therapy receive ibrutinib PO QD on days 1-42 and blinatumomab IV on days 1-28. Treatment repeats every 42 days for up to 3 courses in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE THERAPY: Patients receive ibrutinib PO QD on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Blinatumomab; Drug: Ibrutinib

INTERVENTIONS:
Biological: Blinatumomab — Given IV
  Other Names: Anti-CD19 x Anti-CD3 Bispecific Monoclonal Antibody; Anti-CD19/Anti-CD3 Recombinant Bispecific Monoclonal Antibody MT103; Blincyto; MEDI-538; MT-103
Drug: Ibrutinib — Given PO
  Other Names: BTK Inhibitor PCI-32765; CRA-032765; Imbruvica; PCI-32765

SUMMARY:
This phase II trial studies how well ibrutinib and blinatumomab work in treating patients with B acute lymphoblastic leukemia that has come back or is not responding to treatment. Ibrutinib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Monoclonal antibodies, such as blinatumomab, may interfere with the ability of cancer cells to grow and spread. Giving ibrutinib and blinatumomab may work better in treating patients with relapsed or refractory B acute lymphoblastic leukemia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the efficacy of ibrutinib and blinatumomab in patients with relapsed or refractory B acute lymphoblastic leukemia (B-ALL) as measured by complete response (CR) rate.

SECONDARY OBJECTIVES:

I. To further examine the efficacy and safety of ibrutinib and blinatumomab in patients with relapsed or refractory B-ALL as measured by overall response rate (ORR, defined as CR plus CR with incomplete count recovery [CRi]), relapse free survival (RFS), overall survival (OS), minimal residual disease (MRD) response, proportion of patients bridged to allogeneic hematopoietic cell transplant (allo-HCT), and toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed diagnosis of relapsed or refractory B-cell acute lymphoblastic leukemia/lymphoma with measurable bone marrow lymphoblasts or biopsy-proven extramedullary site measurable by computed tomography (CT) or positron emission tomography (PET)/CT imaging; Philadelphia chromosome-positive (Ph+) B-ALL patients must have failed treatment with at least one second generation tyrosine kinase inhibitor; prior allo-HCT is allowed
* No hematologic parameters for inclusion; transfusion-dependent patients are eligible and platelet counts should be maintained greater than 10,000/mm^3 throughout cycles 1 and 2
* Bilirubin less than or equal to 1.5 x upper limit of normal (ULN) (unless bilirubin rise is due to Gilbert's syndrome or B-ALL or non-hepatic origin)
* Serum aspartate transaminase (aspartate aminotransferase [AST]) or alanine transaminase (alanine aminotransferase [ALT]) less than or equal to 3 x ULN (unless due to B-ALL)
* Estimated creatinine clearance greater than or equal to 30 ml/min (Cockcroft-Gault) or serum creatinine less than or equal to 2 x ULN
* Prothrombin time (PT)/international normalized ratio (INR) =< 1.5 x ULN and partial thromboplastin time (PTT) (activated partial thromboplastin time [aPTT]) =< 1.5 x ULN (unless B-ALL related)
* Karnofsky performance status (KPS) performance status of 60% or greater
* Ability to understand and willingness to sign an informed consent form
* Ability to adhere to the study visit schedule and other protocol requirements
* Female subjects who are of non-reproductive potential (i.e., post-menopausal by history - no menses for >= 1 year; OR history of hysterectomy; OR history of bilateral tubal ligation; OR history of bilateral oophorectomy); female subjects of childbearing potential must have a negative serum or urine pregnancy test within 72 hours prior to the first study drug administration
* Male and female subjects who agree to use both a highly effective methods of birth control (e.g., condoms, implants, injectables, combined oral contraceptives, some intrauterine devices [IUDs], complete abstinence, or sterilized partner) and a barrier method (e.g. condoms, vaginal ring, sponge, etc) during the period of therapy and for 90 days after the last dose of study drug
* Eligibility of patients receiving any medications or substances known to affect or with the potential to affect the activity or pharmacokinetics of ibrutinib or blinatumomab will be determined following review of their case by the investigator

Exclusion Criteria:

* Diagnosis of T acute lymphoblastic leukemia (T-ALL) or Burkitt's leukemia/lymphoma
* Patients with current evidence of active central nervous system (CNS) leukemia
* History of treatment with ibrutinib or blinatumomab
* Investigational therapy, chemotherapy, immunotherapy, radiotherapy, or systemic graft versus host disease (GVHD) therapy within two weeks or five half-lives (whichever is shorter); steroids, hydroxyurea and/or leukapheresis are allowed to control blast count prior to the first dose of study drug
* Prior allo-HCT less than three months from the time of enrollment
* Any active acute GVHD or chronic GVHD greater than grade 1
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to ibrutinib and blinatumomab or other agents used in this study
* Vaccinated with live, attenuated vaccines within 4 weeks of first dose of study drug
* Recent culture-documented infection requiring intravenous antimicrobials that was completed =< 7 days before the first dose of study drug or any uncontrolled active systemic infection; fever of unknown origin is not an exclusion criterion, as this may be disease-related
* Unresolved toxicities from prior anti-cancer therapy, defined as having not resolved to Common Terminology Criteria for Adverse Event (CTCAE, version [v]4.03), grade =< 2, or to the levels dictated in the inclusion/exclusion criteria with the exception of alopecia
* Known bleeding disorders (e.g., von Willebrand's disease) or hemophilia
* History of stroke or intracranial hemorrhage within 6 months prior to enrollment
* Active infection with human immunodeficiency virus (HIV), hepatitis C virus (HCV) or hepatitis B virus (HBV); subjects who are positive for hepatitis B core antibody, hepatitis B surface antigen, or hepatitis C antibody must have a negative polymerase chain reaction (PCR) result before enrollment; those who are PCR positive will be excluded; subjects with HIV must have a CD4 count at or above the institutional lower limit of normal and not taking prohibited CYP3A strong inhibitors
* Major surgery within 4 weeks of first dose of study drug
* Any life-threatening illness, medical condition, or organ system dysfunction, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, active autoimmune disorder, or psychiatric illness/social situations that, in the investigator's opinion, could compromise the subject's safety or put the study outcomes at undue risk; currently active, clinically significant cardiovascular disease, such as uncontrolled arrhythmia or class 3 or 4 congestive heart failure as defined by the New York Heart Association Functional Classification; or a history of myocardial infarction, unstable angina, or acute coronary syndrome within 6 months prior to enrollment
* History of other malignancies, except for malignancy surgically resected (or treated with other modalities) with curative intent, adequately treated in situ carcinoma of the breast or cervix uteri, basal cell carcinoma of the skin or localized squamous cell carcinoma of the skin; malignancy treated with curative intent with no known active disease present for >= 3 years
* Concomitant use of warfarin or other Vitamin K antagonists
* Subjects who received a strong cytochrome P 450 3A (CYP3A) inhibitor within 7 days prior to the first dose of ibrutinib or subjects who require continuous treatment with a strong CYP3A inhibitor
* Currently active, clinically significant hepatic impairment Child-Pugh class B or C according to the Child Pugh classification
* Breastfeeding or pregnant
* Participation in clinical trials with other investigational agents not included in this trial throughout the duration of this trial
* Unwilling or unable to participate in all required study evaluations and procedures or unable to understand the purpose and risks of the study and to provide a signed and dated informed consent form (ICF) and authorization to use protected health information (in accordance with national and local subject privacy regulations)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-06-27 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Rate of CR | Up to 91 days

SECONDARY OUTCOMES:
Incidence of adverse events graded according to the National Cancer Institute CTCAE v4.03 | Up to 6 months
MRD response | Up to 6 months
ORR defined as CR plus CRi assessed by disease-specific response criteria | Up to 6 months
OS | From the time of first study drug administration until the date of progression or death from any cause, assessed for up to 6 months
RFS | Time from CR/CRi until the date of progression or death from any cause, assessed for up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Brian Jonas, Principal Investigator — University of California, Davis
Locations (1):
- University of California Davis Comprehensive Cancer Center, Sacramento, California, United States